CLINICAL TRIAL: NCT02367742
Title: Effect of Two Different Programs of Physical Activity on the Grade of Severity of NAFLD
Brief Title: Effect of Physical Activity on NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Alberto R Osella, MD, PhD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUTRIEPATT
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-02

CONDITIONS: NAFLD
Keywords: Diet; Physical Activity; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endurance Activity (EA) (Other): The subjects have followed a program of endurance (aerobic) activity (EA).
  Interventions: Behavioral: Endurance Activity (EA)
- EA + Resistance Training (RT) (Other): The subjects have followed a program of endurance activity (EA) and resistance training (RT).
  Interventions: Behavioral: EA + Resistance Training (RT)

INTERVENTIONS:
Behavioral: Endurance Activity (EA) — Subjects have followed a program of endurance activity consisting in a 30 minute walk, 5 times/week. Exercise intensity started from the 60% of the maximum heart rate and raised up to the 75%.
  Arms: Endurance Activity (EA)
Behavioral: EA + Resistance Training (RT) — Subjects have followed a program combining endurance activity (EA) and resistance training (RT) consisting in a 60 minute work session, 3 times/week consisting in:
  * Walk (30 minutes): exercise intensity started from the 60% of the maximum heart rate and raised up to the 75%.
  * Musculation (30 minutes): training of the bigger muscle groups (chest, shoulders, arms, abdomen, back, glutei and legs). Exercise intensity started from the 65% of the maximum rated load and raised up to the 75%.
  Arms: EA + Resistance Training (RT)

SUMMARY:
It has been demonstrated the essential role of physical activity in the prevention of overweight and obesity. Nevertheless, the effect of a program of physical activity on the maintenance of body weight in subjects who have previously followed a dietary intervention is still unknown. The aim of this study was to investigate this topic by evaluating the effect of two different programs of physical activity on subjects who have followed a dietary intervention but presented again NAFLD a year after the treatment.

DETAILED DESCRIPTION:
Subjects who were previously enrolled in the trial NUTRIEP and who still have NAFLD a year after the end of the study, were invited to participate in a program of physical activity to assess the effect of endurance and resistance training on weight and NAFLD score. Participants (100 subjects) were randomized and divided into two groups: the first followed a program of endurance activity consisting in a 30 minute walk, 5 times/week; the second followed a program combining the just described aerobic exercise with a resistance training based on 30 minute of musculation involving all the bigger muscles, 3 times/week. The trial lasted six months and subjects underwent liver ultrasonography (to assess NAFLD score), indirect calorimetry, bioimpedenziometry, the measurement of anthropometric variables (body height and weight) and biological parameters (glucose, insulin, cholesterol, HDL cholesterol, triglycerides, GOT, GPT and GGT) at the baseline and at the third and the sixth month. The aim of the study was to estimate the effect of the two different programs of physical activity on NAFLD score. Secondary end-points included: the effect on basal metabolism, the modification of fat mass (FM), lean mass (LM) and muscle mass (MM) and on several biological markers associated with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe NAFLD
* Enrolled in the previous trial called NUTRIEP

Exclusion Criteria:

* Not enrolled in the previous trial called NUTRIEP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in NAFLD score at three and six months | Six months

SECONDARY OUTCOMES:
Change from Baseline in Indirect calorimetry at three and six months | Six months
Percentage Change from Baseline in Bioimpedenziometry at three and six months | Six months
  Percentage reduction in Fat Mass; Percentage increase in Muscle mass

OTHER OUTCOMES:
Height | At baseline
Change from Baseline in Body Weight at three and six months | Six months
Change from Baseline in Systolic blood pressure at three and six months | Six months
Change from Baseline in Diastolic blood pressure at three and six months | Six months
Change from Baseline in Serum Fasting Glucose at three and six months | Six months
Change from Baseline in Serum GOT at three and six months | Six months
Change from Baseline in Serum GPT at three and six months | Six months
Change from Baseline in Serum gamma-GT at three and six months | Six months
Change from Baseline in Serum Cholesterol at three and six months | Six months
Change from Baseline in Serum HDL Cholesterol at three and six months | Six months
Change from Baseline in Serum Triglycerides at three and six months | Six months
Change from Baseline in Serum Insulin at three and six months Insulin | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto R Osella, MD, PhD, Principal Investigator — IRRCS "Saverio De Bellis", Via Turi 27, 70013, Castellana Grotte (Bari), Italy